CLINICAL TRIAL: NCT00546130
Title: Feasibility Study for Multicenter Randomized Controlled Phase III Clinical Trial of Cisplatin + Irinotecan Therapy and Cisplatin + Irinotecan + Krestin Therapy for Extensive-Stage Disease (ED) Small Cell Lung Cancer
Brief Title: Feasibility Study of CDDP + CPT-11 + PSK for Extensive-Stage Disease (ED) Small Cell Lung Cancer
Acronym: RNCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toyama (Other)
Responsible Party: Tatsuhiko Kashii, MD, PhD, Associate Professor, Toyama University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNCLC-01
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-08

CONDITIONS: Small Cell Lung Cancer
Keywords: ED-SCLC; small cell lung cancer; CPT-11; irinotecan hydrochloride; CDDP; cisplatin; PSK; Krestin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Cisplatin; DCM-Dex-CDDP; polysaccharide-K

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Irinotecan hydrochloride + Cisplatin + Krestin Therapy
  Interventions: Drug: Irinotecan hydrochloride; Drug: Cisplatin; Drug: Krestin

INTERVENTIONS:
Drug: Irinotecan hydrochloride — Irinotecan hydrochloride 60 mg/m2, IV (in the vein) on days 1, 8, 15 of each 28 day cycle.
  Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Irinotecan hydrochloride: CPT-11
Drug: Cisplatin — Cisplatin 60 mg/m2, IV (in the vein) on day 1 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Cisplatin: CDDP
Drug: Krestin — Krestin 3,000 mg, PO everyday until progression or unacceptable toxicity develops.
  Other Names: Krestin: PSK

SUMMARY:
The purpose of this study is to examine whether setting test groups of cisplatin + irinotecan + Krestin therapy as first-line treatment and chemotherapy (radiotherapy or radiotherapy + chemotherapy also allowed) combined with Krestin as second-line treatment after exacerbation and comparing with historical control or community control is appropriate as the protocol and regimen for the phase III clinical trial on extensive-stage disease (ED) small cell lung cancer.

DETAILED DESCRIPTION:
To examine whether the following protocol and regimen is appropriate for the phase III clinical trial on extensive-stage disease (ED) small cell lung cancer: set test groups of cisplatin + irinotecan + Krestin therapy as first-line treatment and chemotherapy (radiotherapy or radiotherapy + chemotherapy also allowed) combined with Krestin as second-line treatment after exacerbation, evaluate the efficacy and safety of treatment in a small number of cases, and compare with historical control or community control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven small cell lung cancer
* Patients receiving chemotherapy for the first time
* Patients with no indication for radical radiotherapy or surgical resection
* Patients diagnosed as ED* by full staging [chest X ray, chest C, brain CT or MRI, abdominal CT or abdominal ultrasonography, whole body bone scintigraphy (may be replaced by PET/CT)]

  * ED: Patient with distant metastasis including contralateral hilar lymph node metastasis, but ipsilateral pleural effusion without distant metastasis is excluded.
* Patients with lesions measurable or evaluable by the RECIST criteria
* Patients aged from 20 years to below 75 years
* Patients with preserved organ functions as indicated by the following test values (data obtained within 14 days prior to registration) Hemoglobin: ≥9.0 g/dL White blood cell count: ≥4,000/mm3, ≤12,000 /mm3 Neutrophil count: ≥ 2,000/mm3 Platelet count: ≥100,000 /mm3 GOT, GPT: below 2.5 times the upper limit of normal range for individual facility Total bilirubin: ≤1.5 mg/dL Serum creatinine: below the lower limit of normal range for individual facility Creatinine clearance: ≥ 60mL/min Arterial oxygen tension （PaO2）: ≥60 torr (resting)
* Performance status (PS): 0-1
* Absence of serious concurrent cardiac or pulmonary disease
* Patients expected to survive for at least 3 months
* Patients from whom written informed consent can be obtained

Exclusion Criteria:

* Patients with serious infection and other serious complications (including gastrointestinal bleeding and diarrhea)
* Patients with pleural effusion, ascites, or pericardial effusion that requires treatments including puncture drainage and intracavity administration
* Patients showing definite interstitial pneumonitis or pulmonary fibrosis on plain chest radiograph
* Patients manifesting central nervous system symptoms due to brain metastasis at registration
* Patients with active multiple cancers
* Patients who had undergone bone marrow transplantation
* Patients who had undergone peripheral blood stem cell transplantation
* Patients with a history of definite drug allergy
* Pregnant and nursing patients, patients who may be pregnant or who intend to become pregnant
* Male patients with reproductive capacity who have no intention of contraception during the clinical trial
* Patients with poorly controlled diabetes
* Patients who had been administered Krestin in the past
* Others: patients who are judged by the investigator or subinvestigator to be unsuitable as subject

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | one year

SECONDARY OUTCOMES:
Response rate, Time to treatment failure (TTF), Time to progression (TTP), Progression free survival (PFS), Severity and frequency of toxicity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuhiko Kashii, MD, PhD, Study Chair — Research Network for Chemotherapy of Lung Cancer
Locations (15):
- Japan (15):
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Hiroshima City Hospital, Hiroshima, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa Medical University Hospital, Mukai-awagasaki, Ishikawa-ken
  - Kinkidaigakuigakubu Nara Hospital, Ikoma, Nara
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Osaka Prefectural Medical Center for Respiratory and Allergic Diseases, Habikino, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Kinkidaigakuigakubu Sakai Hospital, Sakai, Osaka
  - NHO Kinki-chuo Chest Medical Center, Sakai, Osaka
  - Osaka Medikal College Hospital, Takatsuki, Osaka
  - Tokyo Medical University Hospital, Tokyo, Tokyo
  - Toyama University Hospital, Toyama, Toyama
  - Toyama Red Cross Hospital, Toyama, Toyama

REFERENCES:
- [Background] Noda K, Nishiwaki Y, Kawahara M, Negoro S, Sugiura T, Yokoyama A, Fukuoka M, Mori K, Watanabe K, Tamura T, Yamamoto S, Saijo N; Japan Clinical Oncology Group. Irinotecan plus cisplatin compared with etoposide plus cisplatin for extensive small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):85-91. doi: 10.1056/NEJMoa003034. PMID 11784874
- [Background] Fisher MD, D'Orazio A. Irinotecan and cisplatin versus etoposide and cisplatin in small-cell lung cancer: JCOG 9511. Clin Lung Cancer. 2000 Aug;2(1):23-4. No abstract available. PMID 14731333
- [Background] Saijo N. Progress in treatment of small-cell lung cancer: role of CPT-11. Br J Cancer. 2003 Dec 15;89(12):2178-83. doi: 10.1038/sj.bjc.6601456. PMID 14676791